CLINICAL TRIAL: NCT01057498
Title: A Phase I Study of Nebulized RNS60 in Adult Healthy Subjects and Patients With Mild to Moderate Asthma.
Brief Title: Safety Study of Nebulized RNS60 to Treat Asthma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01.1.1.H1
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — RNS60

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1a - RNS60 in Healthy Subjects (Experimental): Single dose administration of nebulized RNS60 testing for bronchoconstriction in healthy human subjects.
  Interventions: Drug: RNS60 - single dose
- 1b: RNS60 in Mild Asthmatics (Experimental): Single-dose administration of nebulized RNS60 testing for bronchoconstriction in mild asthmatics.
  Interventions: Drug: RNS60 - single dose
- 2e: RNS60 in mild-to-moderate asthmatics (Experimental): RNS60 in mild-to-moderate asthmatics who are not currently taking a chronic asthma medication.
  Interventions: Drug: RNS60

INTERVENTIONS:
Drug: RNS60 — RNS60, 4ml nebulized twice daily for 15 minutes.
  Arms: 2e: RNS60 in mild-to-moderate asthmatics
Drug: RNS60 - single dose — RNS60, single 4 ml dose nebulized for 15 minutes
  Arms: 1a - RNS60 in Healthy Subjects; 1b: RNS60 in Mild Asthmatics

SUMMARY:
The purpose of this study is two-fold. First, to determine whether nebulized RNS60 is safe in healthy human subjects and in subjects with mild asthma, in a single-dose administration. Second, to determine whether nebulized RNS60 is safe in human subjects with mild-to-moderate asthma over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

For single-dose safety (Groups 1a and 1b):

1. Male or female, aged 18 to 65 years.

2.1. For healthy subjects; clinically considered "healthy" and no diagnosis of asthma.

2.2. For subjects with mild asthma, clinical diagnosis of mild chronic asthma as determined by National Heart, Lung, and Blood Institute's (NHLBI) 2007 guidelines, and who are not regularly using a chronic asthma medication (< 3 doses/week).

3. Subjects must be capable of understanding the purpose and risks of the study and provide written, voluntary informed consent.

4. Women of childbearing potential who have a negative pregnancy test (serum) at the time of study entry.

For multi-dose safety study (Group 2e):

1. Male or female, aged 18 to 65 years.
2. Patients with clinical diagnosis of mild to moderate asthma, as determined by NHLBI 2007 guidelines, who are not already using a chronic asthma medication.
3. Historical documentation of asthma in the patient's medical record.
4. Men and women of reproductive potential who document use of adequate contraception during the study and for 1 month following the last day of treatment (Day 28).
5. Women of childbearing potential who have a negative pregnancy test (serum) at the time of study entry.
6. Subjects, or their legal guardians, must be capable of understanding the purpose and risks of the study and provide written, voluntary informed consent.

Exclusion Criteria (for all groups of the study):

1. With a chronic or acute disease that might interfere with the evaluation of RNS60 therapy.
2. Pregnancy or lactation.
3. Current or prior malignancies (excluding non-melanoma skin carcinoma or carcinoma in situ of the cervix that has been adequately treated).
4. History of infection with human immunodeficiency virus (HIV-1), hepatitis B virus (HBV), or hepatitis C virus (HCV); or Hepatitis A virus (HAV).
5. Infections that require intravenous antibiotic therapy.
6. Significant organ dysfunction, including cardiac, renal, liver, CNS, pulmonary, vascular, gastrointestinal, endocrine, or metabolic (e.g., creatinine ≥ 1.6 mg/dL; ALT or AST ≥ 1.5x the upper limit of normal; history of myocardial infarction, congestive heart failure, or arrhythmias within 6 months prior to study entry).
7. Treatment with a humanized or chimeric antibody therapy within 4 weeks prior to study entry.
8. Treatment with any investigational drugs or therapies within 4 weeks prior to study entry.
9. Any use of antidepressants or other psychiatric medicine in the previous 4 weeks days.
10. Group 1b: Any use of oral, systemic corticosteroids within 2 weeks prior to enrollment. Group 2e: Any use of oral, systemic corticosteroids within 4 weeks prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | 28 days
  Evidence that nebulized RNS60 does not cause bronchoconstriction in subjects with mild-to-moderate asthma, as measured by weekly FEV1 scores over 28 days.

SECONDARY OUTCOMES:
Peak expiratory flow | 28 days
  Evidence that nebulized RNS60 does not cause bronchoconstriction in subjects with mild-to-moderate asthma, as measured by peak expiratory flow measured twice daily over 28 days.
Quality of life | 28 days
  Evidence that nebulized RNS60 does not cause a reduced quality of life in subjects with mild-to-moderate asthma, as measured a weekly quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kari C Nadeau, M.D., Ph.D., Principal Investigator — Stanford University; Richard L Watson, M.D., Study Director — Revalesio Corporation
Locations (2):
- United States (2):
  - West Coast Clinical Trials, Cypress, California
  - Stanford University, Stanford, California